CLINICAL TRIAL: NCT07051538
Title: A Randomized, Double-Blind, Dose-Escalating, Placebo-controlled Phase I Clinical Trial on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Injection or Intravenous Infusion of SHR-1139 Injection in Healthy Chinese Subjects and Multiple Subcutaneous Injections in Patients With Moderate-to-severe Plaque Psoriasis
Brief Title: A Phase I Clinical Trial of Single Subcutaneous Injection or Intravenous Infusion of SHR-1139 Injection in Healthy Chinese Subjects and Multiple Subcutaneous Injections in Patients With Moderate-to-severe Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1139-101
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1139 Injections Group (Experimental)
  Interventions: Drug: SHR-1139 Injections
- SHR-1139 Injections Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-1139 Injections Placebo

INTERVENTIONS:
Drug: SHR-1139 Injections — SHR-1139 injections.
  Arms: SHR-1139 Injections Group
Drug: SHR-1139 Injections Placebo — SHR-1139 injections placebo
  Arms: SHR-1139 Injections Placebo Group

SUMMARY:
This is a clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamic and immunogenicity of SHR-1139 injection in healthy subjects who receive a single subcutaneous injection or intravenous infusion of SHR-1139 injection, and in patients with moderate - to - severe plaque psoriasis who receive multiple subcutaneous injections of SHR-1139 injection.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who fully understand the trial procedures, voluntarily agree to participate, and sign a written informed consent form.
2. Age between 18 and 55 years old (inclusive).
3. Vital signs, physical examinations, laboratory tests, and other assessments are normal or show abnormalities without clinical significance.

Exclusion Criteria:

1. Subjects with any clinical disease in the circulatory, endocrine, nervous, digestive, respiratory, hematological, immunological, psychiatric systems, or metabolic abnormalities; or any other disease that may interfere with trial results.
2. History of malignant tumor.
3. Opportunistic infection within 6 months prior to screening.
4. Acute infection with systemic symptoms requiring systemic intravenous or oral anti-infective treatment within 4 weeks before baseline.
5. Participation in any drug or medical device clinical trial within 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | About 365 days for moderate-to-severe plaque psoriasis subjects
Adverse events (AEs) | About 295 days for healthy subjects.
Serious adverse events (SAEs) | About 295 days for healthy subjects.
Serious adverse events (SAEs) | About 365 days for moderate-to-severe plaque psoriasis subjects.

SECONDARY OUTCOMES:
Serum concentration of SHR-1139 | About 253 days for healthy subjects.
Serum concentration of SHR-1139 | About 365 days for moderate-to-severe plaque psoriasis subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided